CLINICAL TRIAL: NCT01601262
Title: Efficacy and Safety of a Second Series of Low Intensity Extracorporeal Shock Wave Therapy (LI-ESWT) Treatment for Erectile Dysfunction Patients Who Were Partial Responders to the Initial Treatment.
Brief Title: Efficacy & Safety of a 2nd Series of Low Intensity Shock Waves for ED on Partial Responders to First Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0179-12-RMB
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Erectile Dysfunction
Keywords: ED; LI-ESWT
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Experimental)
  Interventions: Device: Low Intensity Extracorporeal Shock waves (Cardiospec 1000)

INTERVENTIONS:
Device: Low Intensity Extracorporeal Shock waves (Cardiospec 1000) — We will apply the cardiospec 1000 unit for LI-ESWL in the penile and inguinal areas, 300 shocks per area, total of 1500 shocks. Full description of treatment series can be seen in the detailed protocol.
  Other Names: Cardiospec 1000

SUMMARY:
Low intensity shock waves (LISW) have been proven in animal studies to induce local growth of new blood vessels. The investigators hypothesized that LISW therapy could improve the symptoms of patients with erectile dysfunction resulting from a problem of blood supply who respond to oral therapy (PDE-5 inhibitors). The current study will check the Efficacy and Safety of a Second Series of LISW Treatment for Erectile Dysfunction Patients Who Were Partial Responders to the Initial Treatment.

DETAILED DESCRIPTION:
The patients will be selected out of the patients with Erectile Dysfunction who received Low intensity shock waves and Were Partial Responders to the treatment.

At the first meeting the patient will receive a full explanation of the study, the potential efficacy and risks. After that the patient will be asked to sign an informed consent form. The patient's general medical condition and any problems related to sexual dysfunction are already known from the previous study he was participating. Also the patient's sexual function is already known by sexual function questionnaires that were filled out in previous study. The criteria for inclusion and exclusion will be reviewed, as well as physical examination. Then shall the patient obtain reporting sexual encounter diaries (SEP) and will be asked to avoid using PDE5i's for a month (washout), if he did not do so of some reason after ending the previous study, then it would be the first visit (Visit 1). At visit 1 The patient will be questioning the sexual function questionnaires without PDE5i's and will pass examination performance Endothelial - FMD, the test takes about 10 minutes, it is not an invasive test (not involved in inserting an instrument or any medication) and is painless. The patient may be asked to also undergo Doppler ultrasound. At the end of visit 1 the patient will begin Series of 12 treatments, in which the subject will be treated twice a week for 3 weeks (6 treatments), then would be discontinuation of the study for 3 weeks, and at the end of this period will be treated twice a week for 3 weeks (6 treatments). Four weeks after the treatment series ends the patient will come for another visit and will be asked to fill in questionnaires and perform the FMD and/or Doppler ultrasound test again. The patient's ED condition will be followed up for a long term after the end of his participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Incomplete response to active treatment (not placebo) on first round but patient is still unsatisfied.
2. Recurring ED (had improved on first round of shock wave therapy but after a certain period of time became clinically worse again) after shock wave therapy.
3. A minimum of two sexual attempts per month.
4. An IIEF-ED domain score ≤ 25 post screening, with or without PDE5i intake according to assessment on final visit of Shockwave previous treatment.
5. A stable heterosexual relationship with the same partner for more than three months

Exclusion Criteria:

1. Subjects that did not respond at all to the first round as well as those that did not respond sufficiently.
2. Any pelvic surgery during the period after the first round.
3. Any unstable medical or psychiatric condition, spinal cord injury, or penile anatomical abnormalities arising during this period .
4. cardiovascular conditions that prevent sexual activity.
5. Recent Use of anti-androgens, or oral or injectable androgens
6. Recent hormonal, neurologic, or psychological pathology

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
IIEF-ED Domain score | 3 months
  Severe ED (6≤IIEF-ED Domain score≤10): an increase of 7 points and above; Moderate ED (11≤IIEF-ED Domain score≤16): an increase of 5 points and above; Mild ED (17≤IIEF-ED Domain score≤25): an increase of 2 points and above.

SECONDARY OUTCOMES:
Rigidity Score Questionaire | 3 months
  An increase of at least 1 point is considered as a treatment success.

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Gruenwald, MD, Principal Investigator — Rambam Health Care Campus; Yoram Vardi, Prof. MD, Study Director — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel